CLINICAL TRIAL: NCT00784823
Title: A Phase I/II Study of Escalating Doses of Bortezomib in Conjunction With High Dose Melphalan as a Conditioning Regimen for Autologous Peripheral Blood Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: Study Combining Bortezomib With High Dose Melphalan to Treat Multiple Myeloma
Acronym: Mel-Vel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 06.05.109B
Record Dates: First submitted 2008-10-31; First posted 2008-11-04 (Estimated); Results first posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan

STUDY DESIGN:
Intervention Model Description: 3 + 3 Dose Escalation
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I Cohort - Bortezomib 1 mg/m2 (Experimental): Bortezomib at 1 mg/m2 on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
  Interventions: Drug: Bortezomib 1 mg/m2; Drug: Melphalan
- Phase I Cohort - Bortezomib 1.3 mg/m2 (Experimental): Bortezomib at 1.3 mg/m2 on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
  Interventions: Drug: Bortezomib 1.3 mg/m2; Drug: Melphalan
- Phase I Cohort - Bortezomib 1.6 mg/m2 (Experimental): Bortezomib at 1.6 mg/m2 on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
  Interventions: Drug: Bortezomib 1.6 mg/m2; Drug: Melphalan
- Phase II Cohort (Experimental): Bortezomib at 1.6 mg/m2 on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
  Interventions: Drug: Bortezomib 1.6 mg/m2; Drug: Melphalan

INTERVENTIONS:
Drug: Bortezomib 1 mg/m2 — * Bortezomib is administered by rapid I.V. push (over 3-5 seconds) via a central or peripheral vein into a flowing saline line
  * Bortezomib will be administered any time on day -4 and 24 hrs after the start of the melphalan infusion on day -1
  * Dosing will be based on actual body weight Patient weight must be measured within seven days of the start of the treatment regimen
  Other Names: Velcade
  Arms: Phase I Cohort - Bortezomib 1 mg/m2
Drug: Bortezomib 1.3 mg/m2 — * Bortezomib is administered by rapid I.V. push (over 3-5 seconds) via a central or peripheral vein into a flowing saline line
  * Bortezomib will be administered any time on day -4 and 24 hrs after the start of the melphalan infusion on day -1
  * Dosing will be based on actual body weight Patient weight must be measured within seven days of the start of the treatment regimen
  Other Names: Velcade
  Arms: Phase I Cohort - Bortezomib 1.3 mg/m2
Drug: Bortezomib 1.6 mg/m2 — * Bortezomib is administered by rapid I.V. push (over 3-5 seconds) via a central or peripheral vein into a flowing saline line
  * Bortezomib will be administered any time on day -4 and 24 hrs after the start of the melphalan infusion on day -1
  * Dosing will be based on actual body weight Patient weight must be measured within seven days of the start of the treatment regimen
  Other Names: Velcade
  Arms: Phase I Cohort - Bortezomib 1.6 mg/m2; Phase II Cohort
Drug: Melphalan — * Melphalan is administered by rapid intravenous infusion via a central or peripheral vein over one hour
  * Melphalan will be dissolved with 10 ml of diluent to a concentration of 5 mg/mL which is then immediately diluted in 0.9% normal saline to a concentration NOT exceeding 0.45 mg/mL prior to administration
  * The final dilution of melphalan is physically and chemically stable for 60 minutes and therefore will be administered within that time period
  * Melphalan will be given as a single dose (not split over 2 or more days)
  * Dosing will be based body surface area calculated using actual body weight
  Other Names: Alkeran

SUMMARY:
The purpose of this study is to determine the tolerance and potential efficacy of combining dose intense melphalan with escalating doses of bortezomib in patients with multiple myeloma undergoing autologous stem cell transplantation.

DETAILED DESCRIPTION:
Multiple myeloma is the second most common hematological malignancy that has affected approximately 40,000 Americans.Conventional chemotherapy has achieved limited control of this disease but studies have reported improved response rates for patients who are treated with dose-intense therapy and autologous hematopoietic stem cell transplantation. This Phase I/II study will investigate the potential of combination therapy of dose-intense melphalan with escalating doses of bortezomib.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of multiple myeloma
2. Show progression of disease after a previous cycle of dose-intense melphalan, or less than 25% decrease in paraprotein measured at 8 weeks after a prior cycle of dose-intense melphalan

   * May have received intervening therapies for disease progression after dose-intense melphalan and enrollment in this protocol
3. Age:18yrs-76yrs at time of melphalan administration
4. Gender: There is no gender restriction
5. Availability of >2x10^6 autologous peripheral blood CD34+ cells/kg or a syngeneic donor meeting eligibility criteria for syngeneic donation

   * Syngeneic transplantation is preferred
   * For patients enrolled in the phase I part of this study, >1x10^6 autologous or syngeneic peripheral blood CD34+ cells/kg remaining in storage as "backup" in case of engraftment failure
6. Recovery from complications of salvage therapy, if administered -

Exclusion Criteria:

1. Diagnosis other than multiple myeloma
2. Chemotherapy or radiotherapy within 28 days of initiating treatment in this study
3. Prior dose-intense therapy within 56 days of initiating treatment in this study
4. Uncontrolled bacterial,viral,fungal or parasitic infections
5. Uncontrolled CNS metastases
6. Known amyloid deposition in heart
7. Organ dysfunction

   * LVEF<40% or cardiac failure not responsive to therapy
   * FVC,FEV1,or DLCO<50% of predicted and/or receiving supplementary continuous oxygen
   * Evidence of hepatic synthetic dysfunction, or total bilirubin>2x or AST>3x ULN
   * Measured creatinine clearance <20ml/min
   * Sensory peripheral neuropathy grade 4
8. Karnofsky score<70% unless a result of bone disease directly caused by myeloma
9. Life expectancy limited by another co-morbid illness
10. History of another malignancy in remission <2yrs (other than basal cell carcinoma)
11. Pregnant (women)or unwilling to use acceptable birth control methods (men or women) for twelve months after treatment
12. Documented hypersensitivity to melphalan or bortezomib or any components of the formulation
13. Patients unable or unwilling to provide consent

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Rowley, MD, Principal Investigator — Director-Blood and Marrow Transplantation Program
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Cohort - Bortezomib Dose 1 mg/m2: Bortezomib at 1 mg/m2 on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
Period: Overall Study
Arm/Group | Phase I Cohort - Bortezomib Dose 1 mg/m2 | Phase I Cohort - Bortezomib 1.3 mg/m2 | Phase I Cohort - Bortezomib 1.6 mg/m2 | Phase II Cohort
Started | 6 | 3 | 3 | 20
Completed | 6 | 3 | 3 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II Cohort: Bortezomib 1.6 mg/m2 on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
- Total: Total of all reporting groups
Arm/Group | Phase I Cohort - Bortezomib Dose 1 mg/m2 | Phase I Cohort - Bortezomib 1.3 mg/m2 | Phase I Cohort - Bortezomib 1.6 mg/m2 | Phase II Cohort | Total
Number analyzed (Participants) | 6 | 3 | 3 | 20 | 32
Age, Continuous [Median (Full Range); unit: years] | 57 [50 to 65] | 63 [55 to 65] | 58 [49 to 61] | 57 [52 to 71] | 57 [49 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 1 | 9 | 17
  Male | 1 | 1 | 2 | 11 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 3 | 20 | 32

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose of Bortezomib (MTD)
Description: The Maximum Tolerated Dose of Bortezomib (MTD) Will be Defined as the Dose Level Prior to That Resulting in Two Out of Six Patients Experiencing a DLT
Time Frame: During dosing of Bortezomib on Day -4 to Day -1 of ASCT
Measure: Number; unit: mg/m2 of bortezomib
Groups:
- Combined Dose Intense Melphalan With Bortezomib (MTD): The purpose of this study is to determine the tolerance and potential efficacy of combining dose intense melphalan with escalating doses of bortezomib in patients with multiple myeloma undergoing autologous stem cell transplantation.
  Combined dose intense Melphalan with maximum tolerated dose of bortezomib (MTD)
  Bortezomib: - Bortezomib is administered by rapid I.V. push (over 3-5 seconds) via a central or peripheral vein into a flowing saline line
  * Bortezomib will be administered any time on day -4 and 24 hrs after the start of the melphalan infusion on day -1
  * Dosing will be based on actual body weight Patient weight must be measured within seven days of the start of the treatment regimen
  Melphalan: - Melphalan is administered by rapid intravenous infusion via a central or peripheral vein over one hour
  * Melphalan will be dissolved with 10 ml of diluent to a concentration of 5 mg/mL which is then immediately diluted in 0.9% normal saline to a concentration NOT exceeding 0.45 mg/mL prior to administration
  * The final dilution of melphalan is physically and chemically stable for 60 minutes and therefore will be administered within that time period
  * Melphalan will be given as a single dose (not split over 2 or more days)
  * Dosing will be based body surface area calculated using actual body weight
Arm/Group | Combined Dose Intense Melphalan With Bortezomib (MTD)
Number analyzed (Participants) | 32
mg/m2 of bortezomib | 1.6

ADVERSE EVENTS:
Description: The limited number of patients limited our ability to analyze groups separately for adverse event reporting. As a result, adverse events were collected irrespective of dose and therefore cannot be separated further.
Groups:
- Phase I Cohort: Bortezomib was dose escalated at 1, 1.3, and 1.6 mg/m2 (3 × 3 design) on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
- Phase II Cohort: Bortezomib 1.6 mg/m2 (3 × 3 design) on days -4 and -1 before transplantation with melphalan 200 mg/m2 given on day -2.
Arm/Group | Phase I Cohort | Phase II Cohort
Serious Adverse Events (participants affected / at risk) | 6/12 | 6/20
Other Adverse Events (participants affected / at risk) | 12/12 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cohort (N=12) | Phase II Cohort (N=20)
Death (General disorders) | 0 | 2
Seizure (Nervous system disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
ICU Admission For Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Engraftment Syndrome (Blood and lymphatic system disorders) | 2 | 0
Guillain-Barre Syndrome (Immune system disorders) | 0 | 1
Neutropenic Fever (Blood and lymphatic system disorders) | 1 | 0
Pulmonary Embolus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Cohort (N=12) | Phase II Cohort (N=20)
Hypotension (Cardiac disorders) | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 6
Diarrhea (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Anorexia (Gastrointestinal disorders) | 4 | 3
Mucositis (Gastrointestinal disorders) | 4 | 4
Esophagitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatic Enzyme Elevations (Gastrointestinal disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 3 | 2
Seizures (Nervous system disorders) | 1 | 0
Fatigue (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Altered Mental Status (Nervous system disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 2
Hypokalemia (Renal and urinary disorders) | 1 | 0
Tumor Lysis Syndrome (Renal and urinary disorders) | 0 | 1
Aspiration Pneumonia (Infections and infestations) | 0 | 2
Fever (Infections and infestations) | 3 | 2
Neutropenic Fever (Infections and infestations) | 3 | 5
Shorness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Humerus Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
C. diff (Infections and infestations) | 1 | 2
Gram-positive bacteremia (Infections and infestations) | 1 | 3
Gram-negative bacteremia (Infections and infestations) | 0 | 1
Polymicrobial sepsis (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Candida Bacteremia (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
The limited number of patients limited our ability to analyze groups separately for adverse event reporting. As a result, adverse events were collected irrespective of dose and therefore cannot be separated further.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes